CLINICAL TRIAL: NCT01160731
Title: A Phase I Dose Finding Study of the Pan-DAC Inhibitor Panobinostat (LBH589) in Combination With Etoposide and Cisplatin in the First Line Treatment of Extensive-Stage Small Cell Lung Cancer - An ICORG In-House Study
Brief Title: Panobinostat, Etoposide, and Cisplatin as First-Line Therapy in Treating Patients With Extensive-Stage Small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-09 ICORG; ICORG-07-09; EUDRACT-2008-003634-21; EU-21047
Record Dates: First submitted 2010-07-09; First posted 2010-07-12 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2012-10

CONDITIONS: Lung Cancer
Keywords: extensive stage small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Cisplatin; etoposide phosphate; Panobinostat

ARMS (1):
- Cisplatin, Etoposide & Panobinostat (Experimental)
  Interventions: Drug: cisplatin; Drug: etoposide phosphate; Drug: panobinostat; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: cisplatin
Drug: etoposide phosphate
Drug: panobinostat
Other: laboratory biomarker analysis
Other: pharmacological study

SUMMARY:
RATIONALE: Panobinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Drugs used in chemotherapy, such as etoposide and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving panobinostat together with etoposide and cisplatin may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of panobinostat when given together with etoposide and cisplatin as first-line therapy in treating patients with extensive-stage small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the maximum-tolerated dose, the recommended dose, and the activity of panobinostat when given in combination with etoposide and cisplatin to patients with extensive-stage small cell lung cancer.

Secondary

* To estimate the time-to-progression, the duration of response, and disease stabilization in these patients.
* To estimate the overall survival of these patients.
* To determine the pharmacokinetic profile of panobinostat in combination with etoposide and cisplatin.
* To assess the overall safety profile of panobinostat in these patients.
* To determine the adverse events in these patients treated with this regimen.
* To assess the quality of life of these patients.

OUTLINE: This is a multicenter, dose-escalation study of panobinostat.

Patients receive chemotherapy comprising cisplatin IV on day 1, etoposide IV on days 1-3, and panobinostat IV over 30 minutes on days 1 and 8. Treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline and then periodically during study treatment and follow up, using questionnaire EQ-5D (Euro QoL).

Blood samples may be collected at baseline and periodically during and after study treatment for pharmacokinetic assessment and biomarker translational studies.

After completion of study treatment, patients are followed up at 4 weeks and then every 3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed small cell lung cancer

  * Extensive-stage disease
* Measurable disease according to RECIST criteria
* No symptomatic brain metastasis or meningeal tumors

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Life expectancy ≥ 6 months
* Absolute neutrophil count > 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10.0 g/dL
* Serum creatinine ≤ 1.5 x upper limit of normal (ULN) OR 24-hour creatinine clearance ≥ to 60 mL/min
* Magnesium, potassium, and phosphorus ≥ the lower limit of normal OR correctable with supplements prior to study treatment
* AST/ALT ≤ 2.5 x ULN (≤ 5.0 x ULN if hepatic metastases are present)
* Serum bilirubin ≤ 1.5 x ULN
* Alkaline phosphatase ≤ 2.5 x ULN OR liver fraction ≤ 2.5 x ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective double contraception (at least 1 barrier method) during and for at least 30 days after completion of study treatment
* No impaired cardiac function, including any one of the following:

  * LVEF < 45% as determined by ECHO
  * Complete left bundle branch block, obligate use of a cardiac pacemaker, congenital long QT syndrome, history or presence of atrial or ventricular tachyarrhythmias, clinically significant resting bradycardia (< 50 beats per minute), QTcF > 480 msec on screening ECG, or right bundle branch block and left anterior hemiblock (bifascicular block)
  * Uncontrolled angina pectoris or acute myocardial infarction within the past 3 months
  * Other clinically significant heart disease (e.g., congestive heart failure, uncontrolled hypertension, history of labile hypertension, or history of poor compliance with an antihypertensive regimen)
* No history of HIV or AIDS-related illness
* No acute or chronic liver or renal disease
* No other concurrent severe and/or uncontrolled medical conditions that could cause unacceptable safety risks or compromise compliance with the protocol, including any of the following:

  * Uncontrolled diabetes
  * Chronic obstructive or chronic restrictive pulmonary disease
  * Active or uncontrolled infection
* No known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to panobinostat, cisplatin, or etoposide
* No hearing impairment that would be a contraindication to the use of cisplatin

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy
* No investigational drug or experimental medications or treatments within the past 30 days or 5 half-lives, whichever is longer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-11; Primary Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated dose (MTD) and recommended dose (RD)
Response rates and toxicity at MTD and RD
Objective response rate according to RECIST criteria

SECONDARY OUTCOMES:
Time to progression according to RECIST criteria
Duration of response or disease stabilization according to RECIST criteria
Overall survival according to RECIST criteria
Effect of the combination regimen on drug pharmacokinetics
Adverse events
Quality of life evaluated by EQ-5D (Euro QoL)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Donnellan, Principal Investigator — Galway University Hospital